CLINICAL TRIAL: NCT02694380
Title: Measuring the Effect of Radiation Therapy on Patient Activity Levels
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Colin E. Champ, MD, Assistant Clinical Professor University of Pittsburgh Radiation Oncology, University of Pittsburgh
Other Study IDs: 15-160
Record Dates: First submitted 2016-01-27; First posted 2016-02-29 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Head and Neck Cancer; Prostate Cancer; Breast Cancer; Lung Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Head and Neck: Subjects with head and neck cancer receiving radiation therapy.
- Prostate: Subjects with prostate cancer receiving radiation therapy.
- Breast: Subjects with breast cancer receiving radiation therapy.
- Lung: Subjects with lung cancer receiving radiation therapy.

SUMMARY:
The goal of this study is to measure the effect of radiation therapy on the activity levels of patients. This will be achieved by tracking their activity levels during a treatment course of radiation therapy.

DETAILED DESCRIPTION:
At the University of Pittsburgh (UPMC) St. Margaret and UPMC Shadyside, in the department of radiation oncology, breast, prostate, head and neck, and lung cancer patients will receive the standard treatment for their cancer and in no way will this study interfere with this treatment. Prior to initiation of radiation, consenting patients will be given Misfit activity tracking devices (accelerometers) to be worn on their wrist to track their activity levels throughout the course radiation therapy. Bracelets will be given to patients by the PI or co-investigators (MDs involved in patient's care) at date of consent and returned at completion of the study. The bracelets will track daily steps taken, calories burned, miles walked, and restful and restless sleep. Again, the purpose of the study is merely to measure the affect radiation therapy has on activity levels of patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Breast, Prostate, Lung or Head and Neck Cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Ability to walk 100 feet without rest
* Signed informed consent

Exclusion Criteria:

* Any other noncutaneous cancer diagnosis under active treatment
* Known metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects are initially referred to the Department of Radiation Oncology for their primary cancer diagnosis. Subjects that fit the diagnosis for this study may be offered participation.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Activity level | up to 15 weeks
  Misfit activity tracking devices (accelerometers) will be worn by patients to track their activity levels 1 day to 4 weeks before radiotherapy, during radiotherapy, and for 1 day to 4 weeks after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, MD, Principal Investigator — UPMC Department of Radiation Oncology
Locations (2):
- United States (2):
  - UPMC St. Margaret Department of Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC Shadyside Department of Radiation Oncology, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No